CLINICAL TRIAL: NCT00236236
Title: CONTAK RENEWAL® Heart Failure Heart Rate Variability Registry
Brief Title: The HF-HRV Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Other Study IDs: CR-CA-022103-H
Record Dates: First submitted 2005-09-02; First posted 2005-10-12 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2005-10

CONDITIONS: Heart Failure; Arrhythmia
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy

SUMMARY:
The Registry will evaluate how HRV Monitor diagnostics change after cardiac resynchronization therapy in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving their first CRT-D
* Patients who sign and date a Patient Informed Consent prior to device implant
* Patients who are available and willing to attend follow-up visits at the study center in which they were enrolled

Exclusion Criteria:

* Patients who are anticipated to receive pacing modes other than DDD or VDD (i.e., chronic atrial fibrillation patients are excluded), or patients who are anticipated to receive adaptive rate therapy
* Patients who are younger than 18 years of age
* Patients whose life expectancy is less than six-months due to other medical conditions
* Patients with or who are likely to receive a tricuspid or other valve prosthesis
* Patients who are currently enrolled in another investigational study that would directly impact the treatment or outcome of the current study
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400
Dates: Start 2003-02; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Kellie Chase, Study Chair — Guidant Corporation